CLINICAL TRIAL: NCT03482986
Title: Role of Dietary Habits in Efficacy of Bariatric Surgery - Study C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017P002526C; R01HL140574 (NIH)
Record Dates: First submitted 2018-03-12; First posted 2018-03-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Bariatric Surgery; Sleeve Gastrectomy; Obesity
Keywords: Diet; Dietary Habits; Weight changes
MeSH Terms: conditions — Obesity; Feeding Behavior; Body Weight Changes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Subject will be advised to follow dietary habits plan A. Since this is a single blind study, the details of the dietary interventions cannot be released during recruitment stage, but will be made public once enrollment closes.
  Interventions: Behavioral: Dietary habits plan
- Group B (Experimental): Subject will be advised to follow dietary habits plan B. Since this is a single blind study, the details of the dietary interventions cannot be released during recruitment stage, but will be made public once enrollment closes.
  Interventions: Behavioral: Dietary habits plan

INTERVENTIONS:
Behavioral: Dietary habits plan — Patients will be given a personalized plan regarding their diet.

SUMMARY:
The purpose of the study is to test how dietary habit interventions affect patients weight loss outcomes after bariatric surgery.

DETAILED DESCRIPTION:
The obesity epidemic is a major public health concern with a significant economic burden in the USA. Bariatric surgery is the most effective and durable weight loss treatment, with long-term cardiometabolic health benefits. Among different types of bariatric procedures, sleeve gastrectomy (SG) has become the most commonly performed in USA. While SG is expected to result in a 50-60% excess weight loss, inter-individual differences in weight loss are large and approximately 25% of patients can be considered poor weight-loss responders who either do not lose a substantial amount of weight or regain the lost weight afterwards. The mechanisms underlying this clinical variation remain unknown and interventions to improve on these outcomes critically lacking. Of interest, altered daily dietary habits are experienced by a substantial proportion of bariatric surgery candidates, raising the question whether such alterations may contribute to inter-individual differences in weight loss success. Therefore, the purpose of the study is to test how dietary habit interventions affect patients weight loss outcomes after bariatric surgery. Since this is a single blind study, the details of the dietary interventions cannot be released during recruitment stage, but will be made public once enrollment closes.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery (sleeve gastrectomy) patients

Exclusion Criteria:

* Insulin-dependent diabetes
* Anemia
* Smoking
* Shift work within the past 1 year
* Drug or alcohol dependency
* Bipolar disorder
* Post traumatic stress disorder (PTSD)

Ages: 22 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Post-intervention change in self-rated hunger | Baseline and 4 weeks (post-intervention)
  Differences in self-rated hunger as measured from the visual analogue scale (VAS; 0-100 score with 0 as ''not at all'' and 100 as ''very much''/''extremely'') questionnaire at baseline and after the intervention

SECONDARY OUTCOMES:
Change in caloric intake | baseline and 4 weeks (post-intervention)
  Difference in caloric intake from baseline to post-intervention
Change in energy expenditure | baseline and 4 weeks (post-intervention)
  resting and postprandial energy expenditure measured by indirect calorimetry
Change in glucose tolerance | baseline and 4 weeks (post-intervention)
  Glucose response to mixed meal test

CONTACTS AND LOCATIONS:
Overall Officials: Frank Scheer, PhD, Principal Investigator — Brigham and Women's Hospital; Ali Tavakkoli, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No